CLINICAL TRIAL: NCT04957693
Title: Effect of Vegan Diet and Lifestyle Changes on the Course and Progression of Indolent Lymphoma During Controlled Waiting Period
Brief Title: Effect of Vegan Diet and Lifestyle Changes on Indolent Lymphoma During Controlled Waiting Period
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: KaMaH - The Center for Health-Promoting Therapies (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0264-18
Record Dates: First submitted 2021-07-05; First posted 2021-07-12 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Indolent Lymphoma
MeSH Terms: interventions — Diet, Vegan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): vegan diet and lifestyle change
  Interventions: Behavioral: vegan diet and lifestyle changes

INTERVENTIONS:
Behavioral: vegan diet and lifestyle changes — vegan diet and lifestyle changes

SUMMARY:
The aim of the present trial is to evaluate the effect of lifestyle changes on the natural history of indolent lymphomas, during the period of watchful waiting. The intervention program is comprised of specifically designed vegan nutrition, physical activity, mostly aerobic, and stress reduction by relaxation and meditation. Outcome results will be followed and analyzed for 3 years, taking into consideration the following parameters - disease burden, specific disease-related symptoms, relevant blood tests, body weight, indicators of well-being. Changes in these parameters will be correlated with the level of compliance and adherence to the intervention program. The results of the trial group of patients will be further compared to the natural history of the disease in a comparable group of patients during their waiting period who were not subject to the above intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patient sex - male and female
* Diagnosis with indolent lymphoma in low-grade lymphoma (follicular lymphoma (FL), marginal zone lymphoma MZL), as assessed by Groupe d'Etude des Lymphomes Folliculaires (GELF) criteria
* Lack of need and non treatable patients at the time of diagnosis
* Existence of detailed medical information about physical activity and dietary habits
* Patients who have signed an informed consent form to participate in the study.

Exclusion Criteria:

* Need for therapeutic intervention
* Administration of chemotherapy and / or monoclonal antibodies or immunomodulatory preparation
* Chronic inflammatory or infectious disease
* Another malignant disease
* Pregnant women, special populations - children and incapacitated of judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | up to 36 months
  Overall Response Rate (ORR) defined as the proportion of patients who achieve complete response (CR) and partial response (PR) determined by PET-CT imaging according to the 2014 Lugano criteria assessing FDG-PET/CT in lymphoma
Partial remission or complete remission | up to 36 months
  Response will be assessed by the revised Lugano classification

SECONDARY OUTCOMES:
Disease Free Survival | up to 36 months
  Disease-free survival defined as the time from the date of the first occurrence of a documented CR to the date of disease progression/ relapse, or death from any cause.
Progression Free Survival | up to 36 months
  The time from the start of treatment to the date of the first documented disease progression or death due to any cause. Based on blood tests, physical exams and Positron Emission Tomography Computed Tomography (PET -CT) Lugano classification

CONTACTS AND LOCATIONS:
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided